CLINICAL TRIAL: NCT05986890
Title: Roux-en-Y Gastric Bypass Versus Loop Gastrojejunostomy for Malignant Gastric Outlet Obstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Gerald P. Wright, Surgical Oncology and Hepatopancreaticobiliary Surgeon, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-433
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Malignant Gastric Outlet Obstruction
Keywords: MGOO; Malignant gastric outlet obstruction; gastric outlet; malignant tumor; proximal bowel obstruction; bowel obstruction
MeSH Terms: conditions — Neoplasms; Intestinal Obstruction | interventions — Anastomosis, Roux-en-Y; Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roux-en-Y Bypass (Other): laparoscopic Roux-en-Y (R-Y) procedure is a well-established procedure, commonly utilized in the setting of bariatric- and gastric cancer surgery. The procedure establishes intestinal continuity that bypasses the distal stomach and duodenum. This is achieved by dividing the jejunum 30-40 cm distal to the ligament of Treitz, bringing the distal end of jejunum up anterior to the transverse colon to be anastomosed to the back wall of the stomach (forming the Roux-limb). The proximal cut end of jejunum then gets anastomosed to the downstream roux-limb (forming the Y-limb). The benefits of this reconstruction include less chance of gastric contents travelling into the afferent limb and similarly, avoiding bile reflux from the afferent limb with associated bile gastritis.
  Interventions: Procedure: Roux-en-Y Bypass
- Gastrojejunostomy (Other): surgical gastrojejunostomy, a procedure dating back to the late 1800's.5 This surgical bypass consists of connecting the stomach to a loop of proximal small bowel, thus bypassing any duodenal or distal gastric obstruction.
  Interventions: Procedure: gastrojejunostomy

INTERVENTIONS:
Procedure: Roux-en-Y Bypass — laparoscopic Roux-en-Y
  Arms: Roux-en-Y Bypass
Procedure: gastrojejunostomy — surgical gastrojejunostomy
  Arms: Gastrojejunostomy

SUMMARY:
This study is intended to investigate whether roux-en-y bypass surgery is superior to conventional loop gastrojejunostomy for Malignant gastric outlet obstruction in terms of tolerance to solid food intake. We hypothesize that roux-en-y bypass will be associated with improved solid food intake in the first 30 days after surgery.

DETAILED DESCRIPTION:
Malignant gastric outlet obstruction is when malignant tumor growth obstructs the gastric outlet at the level of the distal stomach or duodenum, causing food intolerance with nausea and vomiting. Most often, this signifies advanced neoplastic disease with associated poor prognosis for patients. Restoring patients to oral intake is important for palliative purposes. The current standard of care in patients requiring long-term alleviation of symptoms (≥2 months) is performing a loop gastrojejunostomy. This involves creating an intestinal bypass to the site of obstruction in the duodenum or distal stomach. This procedure has long been criticized for its poor resultant function for patients, mainly due to poor tolerance to food intake that include frequent episodes of nausea and vomiting and inability to for solid food intake. The need for a durable solution to malignant gastric outlet obstruction that provides better tolerance to solid food intake is evident. The roux-en-y gastric bypass procedure has been performed for a variety of indications for decades, most commonly for weight loss but also with oncologic resections of the stomach in cases of gastric cancer. Laparoscopic roux-en-y gastric bypass (R-Y bypass) has become the standard for this procedure in experienced hands and has been found to be safe in the short- and long term. The long-term function after R-Y bypass is generally favorable across published literature. No studies exist to compare loop gastrojejunostomy to roux-en-y gastric bypass in patients with malignant gastric outlet obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female aged ≥18 years old.
4. Patients with a diagnosis of malignant gastric outlet obstruction. i. Defined as malignant cancer growth of any organ origin in the area of the distal stomach or duodenum preventing normal gastric emptying as determined by symptoms and cross-sectional imaging studies.

   ii. Symptoms can include abdominal distention, abdominal pain, nausea and vomiting.

   iii. Cross sectional imaging findings can include tumor growth in the area of the distal stomach or duodenum, gastric distention, fluid filled stomach and decompressed bowel distal to obstruction point.
5. Patients deemed to benefit from surgical bypass as opposed to stent placement, by the primary surgeon. This includes assessing participants survival chances and ability to undergo a surgical procedure.
6. Patients in a general health status that permits abdominal surgery under general anesthesia. As determined by primary surgeon and anesthesiologist.

Exclusion Criteria:

1. Patients that have had previous treatment for malignant gastric outlet obstruction.

   a. Including any previous surgery or stent placement for MGOO
2. Patients with MGOO deemed to benefit more from endoscopic stent placement rather than surgery for symptom relief. This assessment will be at treating surgeon's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying as per gastric emptying scintigraphy at 7 days post-operatively. | 7 days post operative
  Results of this study are given as percentage gastric emptying of radioactive (99mTc-SC) nutrients

SECONDARY OUTCOMES:
Gastric emptying study at 30-days | 30 days post operative
  Results of this study are given as percentage gastric emptying of radioactive (99mTc-SC) nutrients
Patient reported daily gastric outlet obstruction scoring system (GOOS) score | 30 days postoperative
  Patients will score each day with the score that reflects the diet that was tolerated that day by the patient. This includes what was able to be ingested without a subsequent vomiting.
Number of Clavien-Dindo grade ≥3 adverse event | 14 days postoperative
Number of patients requiring reoperation for any indication | 30 days postoperative
number of patients with diagnoses of delayed gastric emptying defined as per the International Study Group of Pancreatic Surgery | 30 days postoperative
Time from surgery to death | 100 days postoperative
Improvement of quality of life as measured by short form QOL Questionnaire | measured pre-operatively, at 25-35 days post op and 80-100 days post op
  The short form 36 question QOL questionnaire results in a cumulative score with an increase in score representing a better health-related quality of life
Improvement of quality of life as measured GIQLI | measured pre-operatively, at 25-35 days post op and 80-100 days post op
  The Gastrointestinal quality of life questionnaire results in a cumulative score with an increase in score representing a better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: G. Paul Wright, MD, Principal Investigator — Corewell Health
Locations (1):
- G. Paul Wright, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weaver DW, Wiencek RG, Bouwman DL, Walt AJ. Gastrojejunostomy: is it helpful for patients with pancreatic cancer? Surgery. 1987 Oct;102(4):608-13. PMID 2443991
- [Background] Lillemoe KD, Cameron JL, Hardacre JM, Sohn TA, Sauter PK, Coleman J, Pitt HA, Yeo CJ. Is prophylactic gastrojejunostomy indicated for unresectable periampullary cancer? A prospective randomized trial. Ann Surg. 1999 Sep;230(3):322-8; discussion 328-30. doi: 10.1097/00000658-199909000-00005. PMID 10493479
- [Background] Egrari S, O'Connell TX. Role of prophylactic gastroenterostomy for unresectable pancreatic carcinoma. Am Surg. 1995 Oct;61(10):862-4. PMID 7545358
- [Background] Del Piano M, Ballare M, Montino F, Todesco A, Orsello M, Magnani C, Garello E. Endoscopy or surgery for malignant GI outlet obstruction? Gastrointest Endosc. 2005 Mar;61(3):421-6. doi: 10.1016/s0016-5107(04)02757-9. PMID 15758914
- [Background] ROBINSON JO. The history of gastric surgery. Postgrad Med J. 1960 Dec;36(422):706-13. doi: 10.1136/pgmj.36.422.706. No abstract available. PMID 13742310
- [Background] Doberneck RC, Berndt GA. Delayed gastric emptying after palliative gastrojejunostomy for carcinoma of the pancreas. Arch Surg. 1987 Jul;122(7):827-9. doi: 10.1001/archsurg.1987.01400190093020. PMID 2439057
- [Background] Navarra G, Musolino C, Venneri A, De Marco ML, Bartolotta M. Palliative antecolic isoperistaltic gastrojejunostomy: a randomized controlled trial comparing open and laparoscopic approaches. Surg Endosc. 2006 Dec;20(12):1831-4. doi: 10.1007/s00464-005-0454-5. PMID 17063298
- [Background] Mintziras I, Miligkos M, Wachter S, Manoharan J, Bartsch DK. Palliative surgical bypass is superior to palliative endoscopic stenting in patients with malignant gastric outlet obstruction: systematic review and meta-analysis. Surg Endosc. 2019 Oct;33(10):3153-3164. doi: 10.1007/s00464-019-06955-z. Epub 2019 Jul 22. PMID 31332564
- [Background] Johnsson E, Thune A, Liedman B. Palliation of malignant gastroduodenal obstruction with open surgical bypass or endoscopic stenting: clinical outcome and health economic evaluation. World J Surg. 2004 Aug;28(8):812-7. doi: 10.1007/s00268-004-7329-0. Epub 2004 Aug 3. PMID 15457364
- [Background] Singh SM, Longmire WP Jr, Reber HA. Surgical palliation for pancreatic cancer. The UCLA experience. Ann Surg. 1990 Aug;212(2):132-9. doi: 10.1097/00000658-199008000-00003. PMID 1695834
- [Background] Lucas CE, Ledgerwood AM, Saxe JM, Bender JS, Lucas WF. Antrectomy. A safe and effective bypass for unresectable pancreatic cancer. Arch Surg. 1994 Aug;129(8):795-9. doi: 10.1001/archsurg.1994.01420320017001. PMID 7519417
- [Background] Mittal A, Windsor J, Woodfield J, Casey P, Lane M. Matched study of three methods for palliation of malignant pyloroduodenal obstruction. Br J Surg. 2004 Feb;91(2):205-9. doi: 10.1002/bjs.4396. PMID 14760669
- [Background] Bergamaschi R, Marvik R, Thoresen JE, Ystgaard B, Johnsen G, Myrvold HE. Open versus laparoscopic gastrojejunostomy for palliation in advanced pancreatic cancer. Surg Laparosc Endosc. 1998 Apr;8(2):92-6. PMID 9566559
- [Background] Telford JJ, Carr-Locke DL, Baron TH, Tringali A, Parsons WG, Gabbrielli A, Costamagna G. Palliation of patients with malignant gastric outlet obstruction with the enteral Wallstent: outcomes from a multicenter study. Gastrointest Endosc. 2004 Dec;60(6):916-20. doi: 10.1016/s0016-5107(04)02228-x. PMID 15605006
- [Background] Jeurnink SM, Steyerberg EW, van Hooft JE, van Eijck CH, Schwartz MP, Vleggaar FP, Kuipers EJ, Siersema PD; Dutch SUSTENT Study Group. Surgical gastrojejunostomy or endoscopic stent placement for the palliation of malignant gastric outlet obstruction (SUSTENT study): a multicenter randomized trial. Gastrointest Endosc. 2010 Mar;71(3):490-9. doi: 10.1016/j.gie.2009.09.042. Epub 2009 Dec 8. PMID 20003966
- [Background] Upchurch E, Ragusa M, Cirocchi R. Stent placement versus surgical palliation for adults with malignant gastric outlet obstruction. Cochrane Database Syst Rev. 2018 May 30;5(5):CD012506. doi: 10.1002/14651858.CD012506.pub2. PMID 29845610
- [Background] National Comprehensive Cancer Network. Pancreatic Adenocarcinoma, Version 1.2020. Published 2019. Accessed May 8, 2020. www2.tri-kobe/nccn/guideline/pancreas/english/pancreatic.pdf
- [Background] He L, Zhao Y. Is Roux-en-Y or Billroth-II reconstruction the preferred choice for gastric cancer patients undergoing distal gastrectomy when Billroth I reconstruction is not applicable? A meta-analysis. Medicine (Baltimore). 2019 Nov;98(48):e17093. doi: 10.1097/MD.0000000000017093. PMID 31770192
- [Background] Okuno K, Nakagawa M, Kojima K, Kanemoto E, Gokita K, Tanioka T, Inokuchi M. Long-term functional outcomes of Roux-en-Y versus Billroth I reconstructions after laparoscopic distal gastrectomy for gastric cancer: a propensity-score matching analysis. Surg Endosc. 2018 Nov;32(11):4465-4471. doi: 10.1007/s00464-018-6192-2. Epub 2018 Apr 13. PMID 29654529
- [Background] Nakanishi K, Kanda M, Ito S, Mochizuki Y, Teramoto H, Ishigure K, Murai T, Asada T, Ishiyama A, Matsushita H, Shimizu D, Tanaka C, Kobayashi D, Fujiwara M, Murotani K, Kodera Y. Propensity-score-matched analysis of a multi-institutional dataset to compare postoperative complications between Billroth I and Roux-en-Y reconstructions after distal gastrectomy. Gastric Cancer. 2020 Jul;23(4):734-745. doi: 10.1007/s10120-020-01048-6. Epub 2020 Feb 17. PMID 32065304
- [Background] Edholm D. Early intake of solid food after Roux-en-Y gastric bypass and complications. A cohort study from the Scandinavian Obesity Surgery Registry. Surg Obes Relat Dis. 2018 Sep;14(9):1256-1260. doi: 10.1016/j.soard.2018.05.023. Epub 2018 Jun 6. PMID 30001890
- [Background] Potts JR 3rd, Broughan TA, Hermann RE. Palliative operations for pancreatic carcinoma. Am J Surg. 1990 Jan;159(1):72-7; discussion 77-8. doi: 10.1016/s0002-9610(05)80609-9. PMID 1688485
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Osland E, Yunus RM, Khan S, Alodat T, Memon B, Memon MA. Postoperative Early Major and Minor Complications in Laparoscopic Vertical Sleeve Gastrectomy (LVSG) Versus Laparoscopic Roux-en-Y Gastric Bypass (LRYGB) Procedures: A Meta-Analysis and Systematic Review. Obes Surg. 2016 Oct;26(10):2273-84. doi: 10.1007/s11695-016-2101-8. PMID 26894908
- [Background] Peterli R, Borbely Y, Kern B, Gass M, Peters T, Thurnheer M, Schultes B, Laederach K, Bueter M, Schiesser M. Early results of the Swiss Multicentre Bypass or Sleeve Study (SM-BOSS): a prospective randomized trial comparing laparoscopic sleeve gastrectomy and Roux-en-Y gastric bypass. Ann Surg. 2013 Nov;258(5):690-4; discussion 695. doi: 10.1097/SLA.0b013e3182a67426. PMID 23989054
- [Background] Young MT, Gebhart A, Phelan MJ, Nguyen NT. Use and Outcomes of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Gastric Bypass: Analysis of the American College of Surgeons NSQIP. J Am Coll Surg. 2015 May;220(5):880-5. doi: 10.1016/j.jamcollsurg.2015.01.059. Epub 2015 Feb 16. PMID 25907869
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197